CLINICAL TRIAL: NCT00139919
Title: A Randomized, Double-Blind, Placebo-Controlled, Sequential Panel Study of the Safety and Tolerability of Progressively Decreasing Titration Schedules of Bifeprunox in Subjects With Either Schizophrenia or Bipolar Disorder With an Optional Open-Label 26-Week Extension Study
Brief Title: Progressively Decreasing Titration Schedules of Bifeprunox in Subjects With Schizophrenia or Bipolar Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: H. Lundbeck A/S (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: S154.2.017
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2007-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: Decreasing Titration Study; Schizophrenia; Bipolar; Pharmacokinetic
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — bifeprunox

INTERVENTIONS:
Drug: Bifeprunox

SUMMARY:
This study is to assess the tolerability of bifeprunox with the progressive elimination of titration steps to achieve the shortest tolerated titration dosing to a dose of 40 mg/day in either schizophrenia or bipolar disorder subjects. Study duration is 2 months with an optional open-label 26-week extension study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with the current Diagnosis of Schizophrenia, Bipolar Type I Disorder according to DSM-IV TR criteria
* Age 18 to 55
* Body weight 100-250 lbs
* Be sufficiently stable to allow discontinuation of antipsychotic medication

Exclusion Criteria:

* Acutely psychotic subjects
* Subjects that are acutely manic
* Subjects with a psych diagnosis other than Bipolar Type I Disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2006-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, Orange, California, United States